CLINICAL TRIAL: NCT04302168
Title: Effects of Choline Supplementation on Fetal Growth in Gestational Diabetes Mellitus
Brief Title: Choline Supplementation on Fetal Growth in Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Itamar Futterman, Principal Investigator, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-07-06
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choline Supplement Group (Active Comparator): Choline Supplement 470 mg twice daily for total of 8 weeks.
  Interventions: Dietary Supplement: Choline supplement
- Placebo Group (Placebo Comparator): Placebo pill twice daily for total of 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Choline supplement — Choline 470mg twice daily for 8 weeks.
  Arms: Choline Supplement Group
Dietary Supplement: Placebo — Placebo pill twice daily for 8 weeks
  Arms: Placebo Group

SUMMARY:
Gestational diabetes mellitus (GDM), characterized by maternal high blood sugar, affects up to 15% of pregnancies worldwide. GDM doubles the risk of fetal growth (i.e. macrosomia, large fetus,) which further predisposes the affected fetus to elevated risks of obesity, diabetes and cardiovascular disease later in life. The placenta mediates macrosomia by increasing fat and glucose transport to the fetus during GDM. Effective methods to normalize placental nutrient transport and prevent macrosomia are lacking. Choline is a semi-essential nutrient found in egg yolks, meat, fish and cruciferous vegetables. The demand for this nutrient increases substantially during pregnancy. Previous research demonstrated that maternal choline supplementation (MCS) normalized placental fat and glucose transport as well as fetal growth and fat mass in GDM mice. In this study, the investigators will recruit pregnant women with GDM and randomized them to receive a choline supplement (470mg/day, a dose with demonstrated safety), or a placebo for 8 weeks, starting after gestational week 28. The investigators will determine the effects of choline on fetal growth as well as the influence of choline on placental transport and epigenetic modifications in growth-related genes in the placenta and umbilical cord. Successful completion of this study will provide valuable insights into the use of choline supplement as a modifier of placental macronutrient homeostasis in GDM to improve fetal growth outcomes.

DETAILED DESCRIPTION:
STUDY OBJECTIVES Specific Aim 1: Determine the effect of MCS during pregnancy on birth weight in GDM.

Specific Aim 2: Determine the influence of MCS on macronutrient transport and epigenetic modifications in the placenta and cord blood.

HYPOTHESIS

Aim 1: The investigators hypothesize that the choline group would have lower birth weight and fewer LGA neonates than the non- choline group.

Aim 2: The investigators hypothesize that the choline group would reduce placental transport and increase DNA methylation of metabolic genes.

STUDY DESIGN

Subjects: A convenient sampling methodology will be adopted. The investigators will recruit pregnant women diagnosed with GDM during the second trimester of pregnancy on a rolling basis. Block randomization will be conducted based on treatment methods (i.e. insulin therapy, oral hypoglycemics, or diet only) to randomly assign participants to the intervention and control groups. Recruitment will be conducted using the following methods: (i) study flyers will be posted at the prenatal clinic; (ii) the investigators will identify pregnant women who are potentially eligible by reviewing medical records.

Eligibility Criteria: The inclusion criteria include GDM pregnant women before gestational week 28. GDM is diagnosed with the 2-step process: blood glucose higher than the 140 mg/dL cut-off value after 50 g non-fasting 1-hr and 100 g 3-hr oral glucose challenges. Pregnant women are qualified to participate if they are English- or Spanish- speaking, over 18 years of age, having singleton pregnancy, intending to deliver their babies at the institution and are without any of the conditions listed in the exclusion criteria. Exclusion criteria include pre-existing hyperglycemia, diabetes, cardiovascular conditions and liver disease prior to pregnancy. Patients may choose to participate in the study and not donate a biopsy of their placenta or umbilical cord. Patients who desire stem cell donation or storage will not be able to donate a biopsy of their placenta or umbilical cord. These patients will not be excluded from the primary analysis.

Design and Data Collection Procedures:

All interaction with participants will occur at the delivering hospital while sample analyses will occur at the College where the co-investigator's lab is located. The coordinator for the study, employed by the co-investigators (Brooklyn College), will not access or store data remotely and all data collection and analysis will happen on hospital campus.

The investigators will obtain written informed consent from the pregnant women before study entry. Randomization will be done by pharmacy after patient signs consent. It will be block randomization of 6 patients. After randomization, the investigators will provide the participant in the intervention group with choline supplement pills containing 500 mg of choline bitartrate (235 mg choline, Douglas Lab). The participant will consume 2 pills per day to obtain 470 mg choline for 8 weeks. The recommended intake of choline in the form of Adequate Intake (AI) is 450 mg/d for pregnant women and the Tolerable Upper Intake Level (UL) is 3500 mg/d. Since less than 10% pregnant women reach the AI of choline intake and the upper quartile of choline intake is below 900 mg/d. The dosage that the investigators provide plus the habitual intake of choline in these pregnant women will fall between the AI and UL, i.e. sufficient but not exceeding the limit. The participants in the control group will receive a placebo. Both groups will also receive standard prenatal multivitamins. The investigators will provide the participants with 5 weeks supply of supplements and the investigators will verify their compliance during the time with daily check-off logs of supplement consumption and leftover pill count during their next visit.

The participants will come in for a total of 3 visits at times of routine clinical care. The first visit will be between 24 and 28 weeks of gestation when the investigators enroll the participants, the second visit will be between 28 and 32 weeks of gestation, and the third visit will be between 32 and 36 weeks. The investigators will collect a baseline questionnaire at the first visit (approximately 20 minutes), conduct 3-day dietary recalls after the first visit (approximately 20 minutes, each), and check current weight and collect 20 mL blood samples at all visits. At delivery, the investigators will collect placenta samples and cord blood from the participants.

Baseline questionnaire: The questionnaire includes demographic and medical information such as age, due date, ethnicity, parity, marital status, education level, occupation, household income, medical insurance, substance use, medication use, nutrition supplement, family history of chronic diseases, and self-reported pre-pregnancy weight.

Dietary assessment: Three 24-hr dietary recalls, 2 on weekdays and 1 on a weekend day, will be obtained from each participant by a trained research assistant (RA) via phone calls following the first visits to quantify dietary choline intakes. The multi-pass method of Harnack and colleagues will be used. The RA will record food identification, quantity, ingredient specification, preparation method and enter data into the Nutrition Data System for Research (NDSR) software to analyze choline intake. The RA will also ask participants about their physical activity (PA) during the past 24 hours using the PA recall instrument.

Anthropometric measurements and blood collection: The investigators will measure the participants' weight and height using a medical weighing scale with mechanical height rods during the visits. To minimize food-related concentration differences in plasma biomarkers, participants will be instructed not to consume food for at least 4 hours before their blood draw in the morning. This is a standard recommendation for prenatal visits and is considered as safe. About 20 mL of fasting venous blood will be drawn from each participant during the visits by an investigator. Blood samples will be collected into one EDTA blood collection tube and one serum separator tube and centrifuged to obtain plasma, buffy coat, and serum. Samples will be processed and stored at -80oC at the lab until being used for analytical measurements.

Blood glucose management: The investigators will obtain information about fasting glucose, hemoglobin A1C, medication and insulin therapy from medical charts of the participants.

Birth information and sample collection at delivery: The participants will notify the investigators when they are admitted to the birth center by phone. The investigators will also send them reminders as their due dates are approaching. In addition, the birth center medical staff will be given a list of participant names, thus they will also contact the investigators if a participant checks in when none of the study staff is on site. Once the baby is delivered, the investigators will collect two tubes of cord blood to retrieve serum, plasma, and buffy coat. The investigators will measure the size and weight of the placenta and process the placenta using the following method: full-thickness placental biopsies will be obtained using a 6-mm Keyes punch and stabilized in RNAlater® (for RNA), or frozen in liquid nitrogen (for other purposes). Samples will be transported to the co-investigator's lab for long-term storage at -80C before use.

Dietary intake assessment: As mentioned above, dietary intake data collected from 3-day dietary recalls will be analyzed by the NDSR software. Daily intakes of total choline will be calculated by multiplying the frequency of consumption by the sum of choline derivatives including free choline, phosphatidylcholine (PC), glycerophosphocholine (GPC), phosphocholine, and sphingomyelin of each food item. Daily intakes of betaine (the oxidation product of choline) will be calculated by multiplying consumption frequency and betaine content of each food. Average daily intakes will be calculated as the average daily consumption of total choline and betaine over the 3 days of dietary recalls.

Measurements of choline metabolites: Free choline, betaine and other choline derivatives [e.g. PC, GPC, lysophosphatidylcholine, dimethylglycine, trimethylamine oxide (TMAO)] will be measured in maternal plasma using liquid chromatography (LC)-mass spectrometry (MS) /MS as was conducted in previous studies. To ensure the accuracy and reproducibility of data, stable isotope labeled standards will be used in extraction, all samples will be quantified based on a 6-point standard curve, and each sample will be run in duplicate. Samples with a coefficient of variation (CV) % higher than 5% within run or 10% between run will be rerun.

Specific Aim 2: Determine the influence of MCS on macronutrient transport and epigenetic modifications in the placenta and cord blood. To achieve this aim, the investigators will determine expression of fat and glucose transporters, as well as the upstream regulating pathways AKT/mTOR in placental biopsies from the participants. The investigators will measure the site-specific DNA methylation of key growth and metabolism related genes in the placenta and cord blood.

Analyses of macronutrient transport markers in placental biopsies: To analyze how choline metabolism may be related to placental fat and glucose transport, the investigators will use real-time PCR to quantify mRNA abundance of fat and glucose metabolic genes and transporters, such as glucose transporters GLUT1 and GLUT3, fatty acid metabolism-related genes lipoprotein lipase (LPL), fatty acid translocase (CD36), FATPs, and amino acid transporters SNAT2 and SNAT4. Abundance of respective proteins, as well as phosphorylation of AKT, and mTOR targets 4EBP1 and S6K (indicative of activation of the pathway) will also be measured by western blotting that is routinely conducted in the co-investigator's lab, which includes SDS-PAGE, membrane transfer, incubation with antibodies and visualization with a chemiluminescence imaging system. All primer efficiency and antibody quality will be tested before being used. Both real-time PCR and western blot will be run in triplicate.

Epigenetic regulation of growth and metabolism: the investigators will examine site-specific DNA methylation of genes that are published by previous studies as susceptible to prenatal exposures and mediating long-term growth and metabolic programming of the offspring using bi-sulfite sequencing as was previously conducted. Briefly, genomic DNA will be treated with bisulfite reagent, after which the target genomic region will be amplified by PCR. A MassArray EpiTyper system will be used to quantify methylated sequences. Genes of interest include LEP, SREBP1C, and PPARG which mediates fat metabolism, IGF2 which promotes growth, corticotropin releasing hormone (CRH) which promotes cortisol secretion, and glucocorticoid receptor (GR) which receives cortisol signals.

ELIGIBILITY:
Inclusion Criteria:

* GDM pregnant women before gestational week 28.
* English or Spanish speaking, over 18 years of age
* singleton pregnancy
* intending to deliver their babies at Maimonides Medical Center

Exclusion Criteria:

* pre-existing hyperglycemia
* diabetes
* cardiovascular conditions and liver disease prior to pregnancy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 46 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Birthweight | At time of birth
  Birthweight of neonate

SECONDARY OUTCOMES:
Gene expression of glucose transporters | At time of birth
  Gene expression of glucose transports (GLUT 1 and GLUT3)

CONTACTS AND LOCATIONS:
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrara A. Increasing prevalence of gestational diabetes mellitus: a public health perspective. Diabetes Care. 2007 Jul;30 Suppl 2:S141-6. doi: 10.2337/dc07-s206. No abstract available. PMID 17596462
- [Background] Gillman MW, Rifas-Shiman S, Berkey CS, Field AE, Colditz GA. Maternal gestational diabetes, birth weight, and adolescent obesity. Pediatrics. 2003 Mar;111(3):e221-6. doi: 10.1542/peds.111.3.e221. PMID 12612275
- [Background] Page KA, Romero A, Buchanan TA, Xiang AH. Gestational diabetes mellitus, maternal obesity, and adiposity in offspring. J Pediatr. 2014 Apr;164(4):807-10. doi: 10.1016/j.jpeds.2013.11.063. Epub 2013 Dec 31. PMID 24388326
- [Background] Vohr BR, McGarvey ST, Tucker R. Effects of maternal gestational diabetes on offspring adiposity at 4-7 years of age. Diabetes Care. 1999 Aug;22(8):1284-91. doi: 10.2337/diacare.22.8.1284. PMID 10480772
- [Background] Franks PW, Looker HC, Kobes S, Touger L, Tataranni PA, Hanson RL, Knowler WC. Gestational glucose tolerance and risk of type 2 diabetes in young Pima Indian offspring. Diabetes. 2006 Feb;55(2):460-5. doi: 10.2337/diabetes.55.02.06.db05-0823. PMID 16443781
- [Background] Garcia-Vargas L, Addison SS, Nistala R, Kurukulasuriya D, Sowers JR. Gestational Diabetes and the Offspring: Implications in the Development of the Cardiorenal Metabolic Syndrome in Offspring. Cardiorenal Med. 2012 May;2(2):134-142. doi: 10.1159/000337734. Epub 2012 Apr 12. PMID 22851962
- [Background] Lowe WL Jr, Karban J. Genetics, genomics and metabolomics: new insights into maternal metabolism during pregnancy. Diabet Med. 2014 Mar;31(3):254-62. doi: 10.1111/dme.12352. PMID 24528228
- [Background] Poston L, Bell R, Croker H, Flynn AC, Godfrey KM, Goff L, Hayes L, Khazaezadeh N, Nelson SM, Oteng-Ntim E, Pasupathy D, Patel N, Robson SC, Sandall J, Sanders TA, Sattar N, Seed PT, Wardle J, Whitworth MK, Briley AL; UPBEAT Trial Consortium. Effect of a behavioural intervention in obese pregnant women (the UPBEAT study): a multicentre, randomised controlled trial. Lancet Diabetes Endocrinol. 2015 Oct;3(10):767-77. doi: 10.1016/S2213-8587(15)00227-2. Epub 2015 Jul 9. PMID 26165396
- [Background] Sagedal LR, Overby NC, Bere E, Torstveit MK, Lohne-Seiler H, Smastuen M, Hillesund ER, Henriksen T, Vistad I. Lifestyle intervention to limit gestational weight gain: the Norwegian Fit for Delivery randomised controlled trial. BJOG. 2017 Jan;124(1):97-109. doi: 10.1111/1471-0528.13862. Epub 2016 Jan 14. PMID 26768233
- [Background] Han S, Crowther CA, Middleton P, Heatley E. Different types of dietary advice for women with gestational diabetes mellitus. Cochrane Database Syst Rev. 2013 Mar 28;(3):CD009275. doi: 10.1002/14651858.CD009275.pub2. PMID 23543574
- [Background] Bain E, Crane M, Tieu J, Han S, Crowther CA, Middleton P. Diet and exercise interventions for preventing gestational diabetes mellitus. Cochrane Database Syst Rev. 2015 Apr 12;(4):CD010443. doi: 10.1002/14651858.CD010443.pub2. PMID 25864059
- [Background] Catalano PM, Shankar K. Obesity and pregnancy: mechanisms of short term and long term adverse consequences for mother and child. BMJ. 2017 Feb 8;356:j1. doi: 10.1136/bmj.j1. PMID 28179267
- [Background] Caudill MA. Pre- and postnatal health: evidence of increased choline needs. J Am Diet Assoc. 2010 Aug;110(8):1198-206. doi: 10.1016/j.jada.2010.05.009. PMID 20656095
- [Background] Jiang X, West AA, Caudill MA. Maternal choline supplementation: a nutritional approach for improving offspring health? Trends Endocrinol Metab. 2014 May;25(5):263-73. doi: 10.1016/j.tem.2014.02.001. Epub 2014 Mar 26. PMID 24680198
- [Background] Zeisel SH. Metabolic crosstalk between choline/1-carbon metabolism and energy homeostasis. Clin Chem Lab Med. 2013 Mar 1;51(3):467-75. doi: 10.1515/cclm-2012-0518. PMID 23072856
- [Background] Corbin KD, Zeisel SH. Choline metabolism provides novel insights into nonalcoholic fatty liver disease and its progression. Curr Opin Gastroenterol. 2012 Mar;28(2):159-65. doi: 10.1097/MOG.0b013e32834e7b4b. PMID 22134222
- [Background] Geraghty AA, Lindsay KL, Alberdi G, McAuliffe FM, Gibney ER. Nutrition During Pregnancy Impacts Offspring's Epigenetic Status-Evidence from Human and Animal Studies. Nutr Metab Insights. 2016 Feb 16;8(Suppl 1):41-7. doi: 10.4137/NMI.S29527. eCollection 2015. PMID 26917970
- [Background] Nam J, Greenwald E, Jack-Roberts C, Ajeeb TT, Malysheva OV, Caudill MA, Axen K, Saxena A, Semernina E, Nanobashvili K, Jiang X. Choline prevents fetal overgrowth and normalizes placental fatty acid and glucose metabolism in a mouse model of maternal obesity. J Nutr Biochem. 2017 Nov;49:80-88. doi: 10.1016/j.jnutbio.2017.08.004. Epub 2017 Aug 12. PMID 28915389
- [Background] Jack-Roberts C, Joselit Y, Nanobashvili K, Bretter R, Malysheva OV, Caudill MA, Saxena A, Axen K, Gomaa A, Jiang X. Choline Supplementation Normalizes Fetal Adiposity and Reduces Lipogenic Gene Expression in a Mouse Model of Maternal Obesity. Nutrients. 2017 Aug 18;9(8):899. doi: 10.3390/nu9080899. PMID 28820499
- [Background] Dabelea D. The predisposition to obesity and diabetes in offspring of diabetic mothers. Diabetes Care. 2007 Jul;30 Suppl 2:S169-74. doi: 10.2337/dc07-s211. No abstract available. PMID 17596467
- [Background] Ferrara A, Kahn HS, Quesenberry CP, Riley C, Hedderson MM. An increase in the incidence of gestational diabetes mellitus: Northern California, 1991-2000. Obstet Gynecol. 2004 Mar;103(3):526-33. doi: 10.1097/01.AOG.0000113623.18286.20. PMID 14990417
- [Background] Chen Y, Quick WW, Yang W, Zhang Y, Baldwin A, Moran J, Moore V, Sahai N, Dall TM. Cost of gestational diabetes mellitus in the United States in 2007. Popul Health Manag. 2009 Jun;12(3):165-74. doi: 10.1089/pop.2009.12303. PMID 19534581
- [Background] Kolu P, Raitanen J, Rissanen P, Luoto R. Health care costs associated with gestational diabetes mellitus among high-risk women--results from a randomised trial. BMC Pregnancy Childbirth. 2012 Jul 24;12:71. doi: 10.1186/1471-2393-12-71. PMID 22827919
- [Background] American Diabetes Association. Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S14-80. doi: 10.2337/dc14-S014. No abstract available. PMID 24357209
- [Background] Deputy NP, Sharma AJ, Kim SY, Hinkle SN. Prevalence and characteristics associated with gestational weight gain adequacy. Obstet Gynecol. 2015 Apr;125(4):773-781. doi: 10.1097/AOG.0000000000000739. PMID 25751216
- [Background] Langer O. Management of gestational diabetes: pharmacologic treatment options and glycemic control. Endocrinol Metab Clin North Am. 2006 Mar;35(1):53-78, vi. doi: 10.1016/j.ecl.2005.09.007. No abstract available. PMID 16310642
- [Background] Rosario FJ, Powell TL, Jansson T. Activation of placental insulin and mTOR signaling in a mouse model of maternal obesity associated with fetal overgrowth. Am J Physiol Regul Integr Comp Physiol. 2016 Jan 1;310(1):R87-93. doi: 10.1152/ajpregu.00356.2015. Epub 2015 Oct 21. PMID 26491103
- [Background] Jones HN, Woollett LA, Barbour N, Prasad PD, Powell TL, Jansson T. High-fat diet before and during pregnancy causes marked up-regulation of placental nutrient transport and fetal overgrowth in C57/BL6 mice. FASEB J. 2009 Jan;23(1):271-8. doi: 10.1096/fj.08-116889. Epub 2008 Sep 30. PMID 18827021
- [Background] Brett KE, Ferraro ZM, Yockell-Lelievre J, Gruslin A, Adamo KB. Maternal-fetal nutrient transport in pregnancy pathologies: the role of the placenta. Int J Mol Sci. 2014 Sep 12;15(9):16153-85. doi: 10.3390/ijms150916153. PMID 25222554
- [Background] Sewell MF, Huston-Presley L, Super DM, Catalano P. Increased neonatal fat mass, not lean body mass, is associated with maternal obesity. Am J Obstet Gynecol. 2006 Oct;195(4):1100-3. doi: 10.1016/j.ajog.2006.06.014. Epub 2006 Jul 26. PMID 16875645
- [Background] Hull HR, Thornton JC, Ji Y, Paley C, Rosenn B, Mathews P, Navder K, Yu A, Dorsey K, Gallagher D. Higher infant body fat with excessive gestational weight gain in overweight women. Am J Obstet Gynecol. 2011 Sep;205(3):211.e1-7. doi: 10.1016/j.ajog.2011.04.004. Epub 2011 Apr 14. PMID 21621185
- [Background] Qiao L, Guo Z, Bosco C, Guidotti S, Wang Y, Wang M, Parast M, Schaack J, Hay WW Jr, Moore TR, Shao J. Maternal High-Fat Feeding Increases Placental Lipoprotein Lipase Activity by Reducing SIRT1 Expression in Mice. Diabetes. 2015 Sep;64(9):3111-20. doi: 10.2337/db14-1627. Epub 2015 May 6. PMID 25948680
- [Background] Zeisel SH, Da Costa KA, Franklin PD, Alexander EA, Lamont JT, Sheard NF, Beiser A. Choline, an essential nutrient for humans. FASEB J. 1991 Apr;5(7):2093-8. PMID 2010061
- [Background] Hebbard L, George J. Animal models of nonalcoholic fatty liver disease. Nat Rev Gastroenterol Hepatol. 2011 Jan;8(1):35-44. doi: 10.1038/nrgastro.2010.191. Epub 2010 Nov 30. PMID 21119613
- [Background] Fischer LM, da Costa KA, Kwock L, Galanko J, Zeisel SH. Dietary choline requirements of women: effects of estrogen and genetic variation. Am J Clin Nutr. 2010 Nov;92(5):1113-9. doi: 10.3945/ajcn.2010.30064. Epub 2010 Sep 22. PMID 20861172
- [Background] Raubenheimer PJ, Nyirenda MJ, Walker BR. A choline-deficient diet exacerbates fatty liver but attenuates insulin resistance and glucose intolerance in mice fed a high-fat diet. Diabetes. 2006 Jul;55(7):2015-20. doi: 10.2337/db06-0097. PMID 16804070
- [Background] Fujiki K, Kano F, Shiota K, Murata M. Expression of the peroxisome proliferator activated receptor gamma gene is repressed by DNA methylation in visceral adipose tissue of mouse models of diabetes. BMC Biol. 2009 Jul 10;7:38. doi: 10.1186/1741-7007-7-38. PMID 19589179
- [Background] Cai D, Jia Y, Lu J, Yuan M, Sui S, Song H, Zhao R. Maternal dietary betaine supplementation modifies hepatic expression of cholesterol metabolic genes via epigenetic mechanisms in newborn piglets. Br J Nutr. 2014 Nov 14;112(9):1459-68. doi: 10.1017/S0007114514002402. Epub 2014 Sep 12. PMID 25216241
- [Background] Dimasuay KG, Boeuf P, Powell TL, Jansson T. Placental Responses to Changes in the Maternal Environment Determine Fetal Growth. Front Physiol. 2016 Jan 29;7:12. doi: 10.3389/fphys.2016.00012. eCollection 2016. PMID 26858656
- [Background] Kavitha JV, Rosario FJ, Nijland MJ, McDonald TJ, Wu G, Kanai Y, Powell TL, Nathanielsz PW, Jansson T. Down-regulation of placental mTOR, insulin/IGF-I signaling, and nutrient transporters in response to maternal nutrient restriction in the baboon. FASEB J. 2014 Mar;28(3):1294-305. doi: 10.1096/fj.13-242271. Epub 2013 Dec 13. PMID 24334703
- [Background] Rosario FJ, Kanai Y, Powell TL, Jansson T. Increased placental nutrient transport in a novel mouse model of maternal obesity with fetal overgrowth. Obesity (Silver Spring). 2015 Aug;23(8):1663-70. doi: 10.1002/oby.21165. PMID 26193061
- [Background] Nanobashvili K, Jack-Roberts C, Bretter R, Jones N, Axen K, Saxena A, Blain K, Jiang X. Maternal Choline and Betaine Supplementation Modifies the Placental Response to Hyperglycemia in Mice and Human Trophoblasts. Nutrients. 2018 Oct 15;10(10):1507. doi: 10.3390/nu10101507. PMID 30326592
- [Background] Dhasarathy A, Roemmich JN, Claycombe KJ. Influence of maternal obesity, diet and exercise on epigenetic regulation of adipocytes. Mol Aspects Med. 2017 Apr;54:37-49. doi: 10.1016/j.mam.2016.10.003. Epub 2016 Nov 4. No abstract available. PMID 27825817
- [Background] Heerwagen MJ, Miller MR, Barbour LA, Friedman JE. Maternal obesity and fetal metabolic programming: a fertile epigenetic soil. Am J Physiol Regul Integr Comp Physiol. 2010 Sep;299(3):R711-22. doi: 10.1152/ajpregu.00310.2010. Epub 2010 Jul 14. PMID 20631295
- [Background] Kovacheva VP, Mellott TJ, Davison JM, Wagner N, Lopez-Coviella I, Schnitzler AC, Blusztajn JK. Gestational choline deficiency causes global and Igf2 gene DNA hypermethylation by up-regulation of Dnmt1 expression. J Biol Chem. 2007 Oct 26;282(43):31777-88. doi: 10.1074/jbc.M705539200. Epub 2007 Aug 27. PMID 17724018
- [Background] Jiang X, Yan J, West AA, Perry CA, Malysheva OV, Devapatla S, Pressman E, Vermeylen F, Caudill MA. Maternal choline intake alters the epigenetic state of fetal cortisol-regulating genes in humans. FASEB J. 2012 Aug;26(8):3563-74. doi: 10.1096/fj.12-207894. Epub 2012 May 1. PMID 22549509
- [Background] Wallace TC, Fulgoni VL. Usual Choline Intakes Are Associated with Egg and Protein Food Consumption in the United States. Nutrients. 2017 Aug 5;9(8):839. doi: 10.3390/nu9080839. PMID 28783055
- [Background] Harnack L, Stevens M, Van Heel N, Schakel S, Dwyer JT, Himes J. A computer-based approach for assessing dietary supplement use in conjunction with dietary recalls. J Food Compost Anal. 2008 Feb;21(Suppliment 1):S78-S82. doi: 10.1016/j.jfca.2007.05.004. PMID 19190705
- [Background] Arab L, Tseng CH, Ang A, Jardack P. Validity of a multipass, web-based, 24-hour self-administered recall for assessment of total energy intake in blacks and whites. Am J Epidemiol. 2011 Dec 1;174(11):1256-65. doi: 10.1093/aje/kwr224. Epub 2011 Oct 20. PMID 22021561
- [Background] Timperio A, Salmon J, Crawford D. Validity and reliability of a physical activity recall instrument among overweight and non-overweight men and women. J Sci Med Sport. 2003 Dec;6(4):477-91. doi: 10.1016/s1440-2440(03)80273-6. PMID 14723397
- [Background] Garrison A. Screening, diagnosis, and management of gestational diabetes mellitus. Am Fam Physician. 2015 Apr 1;91(7):460-7. PMID 25884746
- [Background] American Diabetes Association. 13. Management of Diabetes in Pregnancy: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S137-S143. doi: 10.2337/dc18-S013. PMID 29222384
- [Background] Wirfalt AK, Jeffery RW, Elmer PJ. Comparison of food frequency questionnaires: the reduced Block and Willett questionnaires differ in ranking on nutrient intakes. Am J Epidemiol. 1998 Dec 15;148(12):1148-56. doi: 10.1093/oxfordjournals.aje.a009599. PMID 9867258
- [Background] Feskanich D, Sielaff BH, Chong K, Buzzard IM. Computerized collection and analysis of dietary intake information. Comput Methods Programs Biomed. 1989 Sep;30(1):47-57. doi: 10.1016/0169-2607(89)90122-3. PMID 2582746
- [Background] Cho E, Holmes MD, Hankinson SE, Willett WC. Choline and betaine intake and risk of breast cancer among post-menopausal women. Br J Cancer. 2010 Feb 2;102(3):489-94. doi: 10.1038/sj.bjc.6605510. Epub 2010 Jan 5. PMID 20051955
- [Background] Yan J, Jiang X, West AA, Perry CA, Malysheva OV, Brenna JT, Stabler SP, Allen RH, Gregory JF 3rd, Caudill MA. Pregnancy alters choline dynamics: results of a randomized trial using stable isotope methodology in pregnant and nonpregnant women. Am J Clin Nutr. 2013 Dec;98(6):1459-67. doi: 10.3945/ajcn.113.066092. Epub 2013 Oct 16. PMID 24132975
- [Background] Wang Z, Klipfell E, Bennett BJ, Koeth R, Levison BS, Dugar B, Feldstein AE, Britt EB, Fu X, Chung YM, Wu Y, Schauer P, Smith JD, Allayee H, Tang WH, DiDonato JA, Lusis AJ, Hazen SL. Gut flora metabolism of phosphatidylcholine promotes cardiovascular disease. Nature. 2011 Apr 7;472(7341):57-63. doi: 10.1038/nature09922. PMID 21475195
- [Background] Cho CE, Taesuwan S, Malysheva OV, Bender E, Tulchinsky NF, Yan J, Sutter JL, Caudill MA. Trimethylamine-N-oxide (TMAO) response to animal source foods varies among healthy young men and is influenced by their gut microbiota composition: A randomized controlled trial. Mol Nutr Food Res. 2017 Jan;61(1). doi: 10.1002/mnfr.201600324. Epub 2016 Aug 3. PMID 27377678

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/68/NCT04302168/Prot_SAP_000.pdf